CLINICAL TRIAL: NCT03674060
Title: A Dose-block Randomized, Active-controlled, Open-label Clinical Study to Compare Pharmacokinetic Property of SYO-1644 Tab and Nexavar Tab in Healthy Male Volunteers
Brief Title: Study to Compare Pharmacokinetic Property of SYO-1644 Tab. and Nexavar Tab. in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYO-1644
Record Dates: First submitted 2018-09-09; First posted 2018-09-17 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2018-09

CONDITIONS: Healthy, Male
Keywords: Healthy Male Volunteers; Evaluation of the Pharmacokinetic Property; A Dose-block Randomized, Active-controlled, Open-label
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SYO-1644 100mg (Experimental): SYO-1644 tablet, PO, 1 100mg tablet
  Interventions: Drug: SYO-1644
- SYO-1644 150mg (Experimental): SYO-1644 tablet, PO, 1 100mg tablet and 1 50mg tablet
  Interventions: Drug: SYO-1644
- SYO-1644 200mg (Experimental): SYO-1644 tablet, PO, 2 100mg tablet
  Interventions: Drug: SYO-1644
- Nexavar (Active Comparator): Nexavar 200mg/tablet, PO, 1 tablet
  Interventions: Drug: Nexavar tab

INTERVENTIONS:
Drug: SYO-1644 — 100mg: SYO-1644 tablet, PO, 1 100mg tablet
  150mg: SYO-1644 tablet, PO, 1 100mg tablet and 1 50mg tablet
  200mg: SYO-1644 tablet, PO, 2 100mg tablet
  Other Names: SYO-1644 100, 150, 200mg
  Arms: SYO-1644 100mg; SYO-1644 150mg; SYO-1644 200mg
Drug: Nexavar tab — Nexavar 200mg/tablet, PO, 1 tablet
  Other Names: Sorafenib 200mg
  Arms: Nexavar

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics characteristics ,tolerability, and safety after orally administrating SYO-1644 to healthy male volunteers in randomized, active-controlled, open-label clinical study.

DETAILED DESCRIPTION:
After orally administrating SYO-1644 and Nexavar 200 mg to healthy male participants , the safety, tolerability, and pharmacokinetic characteristics are to be compared while testing pharmacokinetic characteristics based on the dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male age between 19 and 50 years old at the time of screening
2. Healthy male more than or equal to 50 kg or less than or equal to 90 kg with BMI of 18~27

   * BMI(kg/m2) = Weight(kg) / {Height(m)}2
3. Agreement with written informed consent

Exclusion Criteria:

1. Participants with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary, psychiatric disorders or history
2. Participants with history of gastrointestinal ulcers, gastritis, gastric ulcer, gastroesophageal reflux disease, Crohn's disease, etc, that may affect the safety and pharmacokinetic evaluation of the test drug, except simple appendectomy and hernia surgery)
3. Participants with hypersensitivity reactions or clinically significant hypersensitivity reactions to drugs including sorafenib and allogeneic drugs, and other drugs (aspirin, antibiotics, etc.)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of pharmacokinetic properties | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 168 hours
  Pharmacokinetics of the AUCt between SYO-1644 and Nexavar cap(200mg)
Evaluation of pharmacokinetic properties | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 168 hours
  Pharmacokinetics of the Cmax between SYO-1644 and Nexavar cap(200mg)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No